CLINICAL TRIAL: NCT05910593
Title: Establishing the Validity and Reliability of a Dexterity Assessment Tool in DCM and Healthy Populations
Brief Title: Establishing the Validity and Reliability of a Dexterity Assessment Tool
Status: Recruiting | Type: Observational
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 123310
Record Dates: First submitted 2023-06-05; First posted 2023-06-20 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Myelopathy Cervical; Cervical Spondylosis; Spinal Cord Compression
MeSH Terms: conditions — Spondylosis; Spinal Cord Compression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Patients diagnosed with degenerative cervical myelopathy; will have dexterity measured once with dexterity tool being tested.
  Interventions: Diagnostic Test: Dexterity Assessment Tool
- Healthy: Healthy volunteers will have their dexterity measured at two time points to perform reliability analysis.
  Interventions: Diagnostic Test: Dexterity Assessment Tool

INTERVENTIONS:
Diagnostic Test: Dexterity Assessment Tool — Measures finger dexterity using pressure sensor pads.

SUMMARY:
Every year, thousands of Canadians are diagnosed with degenerative cervical myelopathy (DCM), a form of non-traumatic injury caused by spinal cord compression in the neck. While DCM causes a range of symptoms, one of the most disabling is loss of hand dexterity. Surgical decompression is standard treatment for DCM, but reduced dexterity often remains.

The investigators have developed a portable, easy-to-use dexterity assessment tool for measuring hand dexterity. Hand function is often assessed using tools incapable of measuring subtle changes in function, limiting a clinician's ability to monitor progression of or recovery from a disease over time. The hope is that if subtle changes in function are identified early, leading to an early DCM diagnosis and treatment, this may prevent patients from experiencing a greater loss of hand function.

The goals of this study are to determine the relationship between dexterity and myelopathy severity, as well as to establish the validity and reliability of the dexterity tool. This will be done by assessing dexterity using the dexterity tool in DCM patients (to determine the relationship between disease severity and dexterity, and measure validity) and healthy participants (to establish reliability).

ELIGIBILITY:
Inclusion criteria for patient participants

* Has been diagnosed with DCM
* Are between the ages of 35 and 75 years
* Has no other neurological disorder Inclusion criteria for healthy participants
* Are between the ages of 35 and 75 years
* Has no neurological disorder

Exclusion criteria for all participants:

• Does not fluently speak and read English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cervical myelopathy patients will be recruited from a neurosurgery clinic.
  Healthy participants will be recruited from individuals who accompany patients to the neurosurgery clinic, in an effort to recruit participants of a similar age to the patient participants.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dexterity measurements using the Dexterity Assessment Tool in patients with cervical myelopathy | Dexterity will be assessed at one time point, when the participant is recruited
  It is anticipated that disease severity will be defined based on the dexterity assessment tool
Correlation between the Dexterity Assessment Tool and the GRASSP-M tool (Graded Redefined Assessment of Strength, Sensation and Prehension-Myelopathy) | Dexterity will be assessed with both tools at one time point, when the participant is recruited
  Concurrent validity will be measured by correlating the Dexterity Assessment Tool with another validated tool, the GRASSP-M
Correlation of dexterity measurements in healthy participants using the Dexterity Assessment Tool to measure inter-rater reliability | Dexterity will be assessed in healthy participants at one time point, when the participant is recruited.
  Inter-rater reliability will be assessed by measuring dexterity in healthy participants with two testers administering the tool one hour apart, and correlating the values from the two testers.
Correlation of dexterity measurements in healthy participants using the Dexterity Assessment Tool to measure test-retest reliability | Dexterity well be assessed in healthy participants at two time points, once when the participant is recruited, and once one week later.
  Test-retest reliability will be assessed by measuring dexterity in healthy participants at two time points, one week apart. The data from the two time points will be correlated to determine reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- LHSC - University Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No